CLINICAL TRIAL: NCT04077333
Title: Minimal Invasive Surfactant Administration to Treat Neonatal Respiratory Distress Syndrome: a Multicenter Clinical Study in China
Brief Title: MISA to NRDS：a Multicenter Study in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Han Tongyan, Vice Director of Pediatrics Department, Principal Investigator, Clinical Associated Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2017160
Record Dates: First submitted 2019-07-10; First posted 2019-09-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Bronchopulmonary Dysplasia; Patent Ductus Arteriosus; Intraventricular Hemorrhage; Necrotizing Enterocolitis; Periventricular Leukomalacia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Ductus Arteriosus, Patent; Enterocolitis, Necrotizing; Leukomalacia, Periventricular

STUDY DESIGN:
Intervention Model Description: A randomized, clinical, parallel-group study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MISA group (Experimental): minimal invasive surfactant administration group
  Interventions: Procedure: Minimal Invasive surfactant administration
- EISA group (No Intervention): conventional treatment: endotracheal intubation surfactant administration group

INTERVENTIONS:
Procedure: Minimal Invasive surfactant administration — Participants enrolled spontaneously breathing preterm infants born between 26.1 and 31.9 weeks' gestational age with signs of respiratory distress syndrome. Preterm infants of the MISA (Minimal invasive surfactant administration) group were assigned to receive surfactant (Calf pulmonary surfactant, Double-Crane Pharmaceutical Co., China) via a 5Fr nasogastric tube with an ophthalmic surgery straight forceps during CPAP/NIPPV-assisted spontaneous breathing.
  Arms: MISA group

SUMMARY:
BACKGROUND Treatment of neonatal respiratory distress syndrome with exogenous surfactant and mechanical ventilation made millions of preterm infants survived in neonatal intensive care unit (NICU). Endotracheal intubation surfactant administration is related to invasive intubation and short periods of positive pressure ventilation and implies the risk of lung injury. Continuous positive airway pressure (CPAP) or NIPPV (Non-invasive positive pressure ventilation) with surfactant but without intubation may work synergistically. This randomized trial investigated a minimal invasive surfactant administration (MISA). To test the hypothesis that MISA increases survival without bronchopulmonary dysplasia (BPD) at 36 weeks' gestational age in very low birth weight infants.

DESIGN, SETTING, AND PARTICIPANTS The Minimal Invasive Surfactant Administration (MISA) was a multicenter, randomized, clinical, parallel-group study conducted between July 1st, 2017, and November 30, 2018, in 8 level III neonatal intensive care units in Beijing, Tianjin, and Hebei province, China. The final follow-up date was March 30, 2019. Participants enrolled spontaneously breathing preterm infants born between 26.1 and 31.9 weeks' gestational age with signs of respiratory distress syndrome. In an intention-to-treat design, infants were randomly assigned to receive surfactant (Calf pulmonary surfactant, Double-Crane Pharmaceutical Co., China) either via a 5Fr nasogastric tube during CPAP/NIPPV-assisted spontaneous breathing (minimal invasive surfactant administration group, MISA group) or after conventional endotracheal intubation during mechanical ventilation (endotracheal intubation surfactant administration group, EISA group).

INTERVENTION MISA via a 5Fr nasogastric tube with an ophthalmic surgery straight forceps.

ELIGIBILITY:
Inclusion Criteria:

1. preterm infants born before 32 weeks gestational age
2. spontaneously breathing receiving continuous positive airway pressure (CPAP) or NIPPV (Non-invasive positive pressure ventilation) without intubation
3. clinical diagnosis of respiratory distress syndrome.

Exclusion Criteria:

1. with obvious malformations
2. with asphyxia requiring intubation during resuscitation
3. need endotracheal intubation or mechanical ventilation before surfactant administration.

Ages: 1 Hour to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of bronchopulmonary dysplasia (BPD) | At 36 weeks'gestational age
  Number of very low birth weight preterm infants with BPD

SECONDARY OUTCOMES:
Incidence of major complications | Through study completion and up to corrected three months
  Number of very low birth weight preterm infants diagnosed with major complications (i.e.patent ductus arteriosus,pulmonary hemorrhage, intraventricular hemorrhage, periventricular leukomalacia, necrotizing enterocolitis, and retinopathy of prematurity）

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Tong, Master, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No